CLINICAL TRIAL: NCT00445757
Title: Evaluation of a Radio-Surgical Approach for the Treatment of Kidney Tumors
Brief Title: Stereotactic Radiation Therapy in Treating Patients With Kidney Tumors
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: slow accrual
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE5806; P30CA043703 (NIH); CASE5806 (Other: Case Comprehensive Cancer Center)
Record Dates: First submitted 2007-03-07; First posted 2007-03-09 (Estimated); Last update posted 2012-03-20 (Estimated); Status verified 2012-03

CONDITIONS: Kidney Cancer
Keywords: stage I renal cell cancer; stage II renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: conventional surgery — Two months after completion of radiotherapy, patients undergo preoperative assessment of tumor response followed by partial nephrectomy.
Radiation: stereotactic radiosurgery — Patients undergo stereotactic radiotherapy to 1 tumor. Cohorts of 4-8 patients receive escalating doses of radiotherapy twice daily for 2 days until the maximum tolerated dose (MTD) or upper limit is reached.

SUMMARY:
RATIONALE: Stereotactic radiation therapy may be able to send x-rays directly to the tumor and cause less damage to normal tissue. Giving stereotactic radiation therapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

PURPOSE: This phase I trial is studying the side effects and best dose of stereotactic radiation therapy in treating patients with kidney tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of radiation in patients undergoing stereotactic radiotherapy for renal tumors.
* Determine radiotherapy-associated toxicity in these patients.

Secondary

* Determine preoperative pathologic response to this regimen in these patients.

OUTLINE: This is a dose-escalation study of radiotherapy.

* Radiotherapy: Patients undergo stereotactic radiotherapy to 1 tumor. Cohorts of 4-8 patients receive escalating doses of radiotherapy twice daily for 2 days until the maximum tolerated dose (MTD) or upper limit is reached. The MTD is defined as the dose preceding that at which at least 2 of 4 or 3 of 8 patients experience dose-limiting toxicity (DLT). DLT is assessed at 4 and 8 weeks after radiotherapy.
* Surgery: Two months after completion of radiotherapy, patients undergo preoperative assessment of tumor response followed by partial nephrectomy.

After completion of study therapy, patients are followed periodically for at least 2 years.

PROJECTED ACCRUAL: A total of 20 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Radiologically confirmed renal tumor

  * At least 4 cm in greatest dimension
* No clinically, radiologically, or pathologically involved lymph nodes
* No distant metastases

PATIENT CHARACTERISTICS:

* Karnofsky performance status 70-100%
* Negative pregnancy test
* Fertile patients must use effective contraception
* Medically eligible for tumor resection
* No major medical condition or psychiatric illness that would preclude study compliance
* No active connective tissue disease, such as lupus or dermatomyositis
* No active Crohn's disease or active ulcerative colitis

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy
* No prior abdominal or pelvic radiotherapy
* No prior cryosurgery
* No prior radiofrequency ablation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-01; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of radiation | DLT is assessed at 4 and 8 weeks after radiotherapy
Radiotherapy-associated toxicity | DLT is assessed at 4 and 8 weeks after radiotherapy

SECONDARY OUTCOMES:
Disease-free survival | follow-up will be done at 1 month, 6 12, 18 and 24 months post surgery
Time to local progression | follow-up will be done at 1 month, 6 12, 18 and 24 months post surgery
Time to distant failure | follow-up will be done at 1 month, 6 12, 18 and 24 months post surgery
Survival | follow-up will be done at 1 month, 6 12, 18 and 24 months post surgery
Disease-specific survival | follow-up will be done at 1 month, 6 12, 18 and 24 months post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Lee E. Ponsky, MD, Principal Investigator — Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Locations (1):
- Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States